CLINICAL TRIAL: NCT06582303
Title: Analysis of the Effectiveness of Visual Training in Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Science and Technology, Pakistan (Other)
Responsible Party: Principal Investigator, Dr. Asim Waris, Dr, National University of Science and Technology, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMES/REC/22/027
Record Dates: First submitted 2024-08-24; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Stroke, Subacute
Keywords: VR games; Visual feedback; Intervention; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Subacute stroke patients were randomly assigned to the experimental group and the control group. The experimental group received a VR hand game intervention along with conventional physical therapy, while the control group only received conventional physical therapy. Each patient's therapy consists of 24 sessions, with each session lasting 4 days per week for a total duration of 6 weeks. The VR intervention consists of four games that utilize a virtual reality device and are controlled by affected hand movements such as flexion/extension, close/open, supination/pronation, and pinch. The control group and experimental groups received conventional physical therapy, which consists of range of motion, stretching, resistance, and strengthening exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Virtual reality intervention plus conventional physical therapy (Experimental): The experimental group initially got VR intervention by playing all four easy-level games twice for three minutes each during the first and second weeks. This group again underwent VR intervention, playing all four same games with a difficulty level of twice 5 min duration for the third, fourth, fifth, and sixth weeks. The experimental group had an intervention of 24 sessions, lasting 4 days/week for a total of 6 weeks. During the first two weeks, patients received 24 minutes of VR hand games and 24 minutes of therapy sessions per day and for the next four weeks, this group received 40 minutes of VR hand games and 40 minutes of conventional therapy session per day. This group received conventional physical therapy that consists of range of motion, stretching, resistance, and strengthening exercises. At follow-up of two weeks this group only received conventional physical therapy.
  Interventions: Device: Virtual reality Game intervention plus conventional physical therapy
- Control Group: Conventional physical therapy (Active Comparator): The control group received conventional physical therapy, which consists of range of motion, stretching, resistance, and strengthening exercises. The CPT group had a conventional intervention of 24 sessions, lasting 4 days per week for a total of 6 weeks. The CPT group was given 48 minutes of conventional physical therapy sessions per day for weeks 1 and 2, followed by 80 minutes of conventional physical therapy sessions per day for the next 4 weeks. At a follow-up of two weeks, this group also received conventional physical therapy.
  Interventions: Device: Conventional Physical Therapy

INTERVENTIONS:
Device: Virtual reality Game intervention plus conventional physical therapy — The experimental group initially got VR intervention by playing all four easy-level games named hitting a rolling ball, grasping a balloon, swapping hands, and gripping twice for three minutes each during the first and second weeks. This group again underwent VR intervention by playing all four same games with a difficulty level twice 5 min duration for the third, fourth, fifth, and sixth weeks. The experimental group had an intervention of 24 sessions, lasting 4 days/week for a total of 6 weeks. During the first two weeks, patients received 24 minutes of VR hand games and 24 minutes of therapy sessions per day and for the next four weeks, this group received 40 minutes of VR hand games and 40 minutes of conventional therapy session per day. This group received conventional physical therapy that consists of range of motion, stretching, resistance, and strengthening exercises. At follow-up of two weeks this group only received conventional physical therapy.
  Other Names: VRGI+CPT
  Arms: Experimental Group: Virtual reality intervention plus conventional physical therapy
Device: Conventional Physical Therapy — The control group received conventional physical therapy, which consists of range of motion, stretching, resistance, and strengthening exercises by using powerweb, thera putty, and occupational therapy equipment. The CPT group had a conventional intervention of 24 sessions, lasting 4 days/week for a total of 6 weeks. The CPT group was given 48 minutes of conventional physical therapy sessions per day for weeks 1 and 2 followed by 80 minutes of conventional physical therapy sessions per day for the next 4 weeks. At follow-up of two weeks, this group also received conventional physical therapy.
  Other Names: CPT
  Arms: Control Group: Conventional physical therapy

SUMMARY:
The study was a randomized control trial conducted to determine whether VR games incorporated with cognitive engagement within visual training feedback are feasible intervention options in stroke rehabilitation. An investigation has been conducted to assess the efficacy of virtual reality games that enhance hand motor functions to attain long-lasting improvements. Patients were randomly assigned to the experimental and control groups. Each patient's therapy consists of 24 sessions, with each session lasting 4 days per week, for a total duration of 6 weeks. Developed four VR-based hand games that include hitting a rolling ball, grasping a balloon, swapping hands, and gripping a pencil.

DETAILED DESCRIPTION:
The field of stroke rehabilitation frequently faces limitations in therapies and struggles to achieve long-lasting improvements in hand motor function. The integration of fully immersive virtual reality (VR) games with visual training feedback significantly improves the efficacy of stroke rehabilitation. Virtual reality (VR) games that incorporate repetitive and particular tasks stimulate the gradual activation of brain pathways linked to motor activities. VR research has the potential to enhance VR intervention games by combining cognitive engagement with visual feedback.

The objective of this study was to develop and evaluate virtual reality games that utilize an approach of cognitive engagement within visual feedback in order to enhance hand-motor capabilities. The study utilized completely immersive virtual reality (VR) games specifically designed for subacute stroke patients. The implementation of fully immersive virtual reality (VR) games as an intervention proved to be highly effective in significantly maintaining the motor recovery of patients who had experienced a stroke in the subacute phase. Stroke patients exhibited enhanced dexterity, heightened range of motion, greater hand strength, and improved grip.

Developed VR games utilize a virtual reality device and are designed to be controlled by hand movements such as flexion/extension, close/open, supination/pronation, and pinch. Patients were randomly assigned to the experimental and control groups. The experimental group received a VR hand game intervention with conventional physical therapy, while the control group only received conventional physical therapy. Each patient's therapy consists of 24 sessions, with each session lasting 4 days per week for a total duration of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Montreal Cognitive Assessment (MOCA ≥ 21)
* Modified Ashworth Scale (MAS< 4)
* Fugl-Meyer Assessment (FMA between 25 and 55)
* Age ≥ 18 years
* Stroke patient type (Subacute patients)

Exclusion Criteria:

* Wrist Impairments
* Contractures
* Patients with vestibular issues
* Permanent external fixation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment-Upper Extremity (FMA-UE) | Baseline, 4th week, 6th week, and 9th week (follow-up)
  The Fugl-Meyer Assessment-Upper Extremity subscale was employed to examine the motor function restoration in the upper extremity of stroke patients following interventions. The Fugl-Meyer Assessment-Upper Extremity consists of 33 items that assess motor function, with a scoring range of 0-66, The minimum score 0 represents severe impairment, and maximum score 66 represents normal motor function. Higher scores indicate better motor function.
Action Research Arm Test (ARAT) | Baseline, 4th week, 6th week, and 9th week (follow-up)
  The Action Research Arm Test is utilized to examine the functional capabilities of stroke patients upper extremities, specifically in terms of reaching, gripping, pinching, and overall movement tasks. Each item is allocated a rating score of 4 points, with the potential total values ranging from 0 to 57. The minimum score 0 represents severe impairment, and the maximum score 57 represents normal upper extremity function. Higher scores on the Action Research Arm Test indicate better functional capabilities of the upper extremities.
Box and Block Test (BBT) | Baseline, 4th week, 6th week, and 9th week (follow-up)
  The BBT evaluated the manual dexterity of individuals who had suffered a stroke. During this assessment, participants are required to transfer blocks from one container to another within a one-minute time limit.
Correlation between electromyography signal features and clinical outcomes | Baseline, 4th week, 6th week, and 9th week (follow-up)
  Electromyography signals are obtained in order to evaluate the electrical activity generated by muscles. Electromyography was utilized for the objective assessment of the effectiveness of immersive VR-based hand games. The objective assessment includes the evaluation of the correlation between electromyography signal features and clinical outcomes, which includes the Fugl-Meyer Assessment-Upper Extremity, Action Research Arm Test, and Box and Block Test.
Movement performance | Baseline, 4th week, 6th week, and 9th week (follow-up)
  The weekly movement performance was evaluated by machine learning algorithms that include k-nearest neighbors, random forest, and support vector machine classifiers on the electromyography signals of stroke patients.

SECONDARY OUTCOMES:
Modified Barthel Index (MBI) | Baseline and 9th week (follow-up)
  The Modified Barthel Index assesses an individual's ability to perform both practical and routine tasks independently. The Modified Barthel Index consists of 10 items, each scored based on the level of assistance required or the level of autonomy demonstrated by the patient. The total score ranges from a minimum of 0 to a maximum of 20. Lower scores indicate greater dependence, with scores below 10 typically representing severe disability and scores below 15 usually indicating moderate disability. Moreover, higher scores reflect greater independence in performing daily activities.
Stroke-Specific Quality of Life (SSQOL) | Baseline and 9th week (follow-up)
  The Stroke-Specific Quality of Life measure was used to assess the health-related quality of life of stroke survivors. The Stroke-Specific Quality of Life scale consists of 49 comprehensive items that evaluate various aspects of quality of life based on the patient's current state. The total score ranges from a minimum of 49 to a maximum of 245. Lower scores indicate poorer health-related quality of life, and higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Asim Waris, PhD, Study Chair — National University of Sciences and Technology (NUST), Islamabad, Pakistan
Locations (1):
- Physiotherapy Department, Holy Family Hospital., Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bae S, Park HS. Development of Immersive Virtual Reality-Based Hand Rehabilitation System Using a Gesture-Controlled Rhythm Game With Vibrotactile Feedback: An fNIRS Pilot Study. IEEE Trans Neural Syst Rehabil Eng. 2023;31:3732-3743. doi: 10.1109/TNSRE.2023.3312336. Epub 2023 Sep 28. PMID 37669214
- [Background] Fregna G, Schincaglia N, Baroni A, Straudi S, Casile A. A novel immersive virtual reality environment for the motor rehabilitation of stroke patients: A feasibility study. Front Robot AI. 2022 Aug 29;9:906424. doi: 10.3389/frobt.2022.906424. eCollection 2022. PMID 36105763
- [Background] Lange B, Koenig S, Chang CY, McConnell E, Suma E, Bolas M, Rizzo A. Designing informed game-based rehabilitation tasks leveraging advances in virtual reality. Disabil Rehabil. 2012;34(22):1863-70. doi: 10.3109/09638288.2012.670029. Epub 2012 Apr 12. PMID 22494437
- [Background] Hernandez A, Bubyr L, Archambault PS, Higgins J, Levin MF, Kairy D. Virtual Reality-Based Rehabilitation as a Feasible and Engaging Tool for the Management of Chronic Poststroke Upper-Extremity Function Recovery: Randomized Controlled Trial. JMIR Serious Games. 2022 Sep 27;10(3):e37506. doi: 10.2196/37506. PMID 36166289
- [Background] Huang J, Lin M, Fu J, Sun Y, Fang Q. An Immersive Motor Imagery Training System for Post-Stroke Rehabilitation Combining VR and EMG-based Real-Time Feedback. Annu Int Conf IEEE Eng Med Biol Soc. 2021 Nov;2021:7590-7593. doi: 10.1109/EMBC46164.2021.9629767. PMID 34892847
- [Result] Amin F, Waris A, Syed S, Amjad I, Umar M, Iqbal J, Omer Gilani S. Effectiveness of Immersive Virtual Reality-Based Hand Rehabilitation Games for Improving Hand Motor Functions in Subacute Stroke Patients. IEEE Trans Neural Syst Rehabil Eng. 2024;32:2060-2069. doi: 10.1109/TNSRE.2024.3405852. Epub 2024 May 30. PMID 38801680